CLINICAL TRIAL: NCT06802133
Title: Monitoring the Use of Collagen Dural Regeneration Matrix (DuraMatrix-Onlay Plus) in the Postmarket Phase.
Brief Title: Post-Market Clinical Investigation Plan- Collagen Dural Regeneration Matrix (DuraMatrix-Onlay Plus)
Status: Recruiting | Type: Observational
Sponsor: Collagen Matrix (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP.057_DMOP
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Repair of Dura Mater

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: Post Market Study — Prospective case series without a concurrent comparator group.

SUMMARY:
Monitoring the Use of Collagen Dural Regeneration Matrix (DuraMatrix-Onlay Plus) in the Postmarket Phase.

DETAILED DESCRIPTION:
A prospective, post-market, open label clinical study at a maximum of 8 sites, with an enrollment of 118 subjects. The primary endpoint of the study will be the rate of revision surgery. The presence of adverse events will be evaluated at each follow-up time point i.e. CSF leak, infection and Pseudomeningocele. Patients will have a follow-up evaluation at least at 8 weeks post initial surgery date (which align with the approximate resorption time of the device) where possible and as deemed necessary by a clinician.

No original patient records or personal identifying information will be disclosed to Collagen Matrix.

ELIGIBILITY:
Inclusion Criteria:

* The general population will be included in the study where a dura substitute is required for the repair of dura mater.

Exclusion Criteria:

* Patients that have conditions which are contraindicated per the instructions for use (IFU) would be excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The general population will be included in the study where a dura substitute is required for the repair of dura mater
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Revision Surgery | 8 weeks
  Adequate healing of dural defects without need for a revision surgery or second intervention

SECONDARY OUTCOMES:
Rate of Adverse events | 8 weeks
  Rate of product-related adverse events or complications

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Augusta University, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts